CLINICAL TRIAL: NCT07056777
Title: A Phase Ib/IIa Clinical Trial Evaluating the Preliminary Efficacy and Safety of DR30206 in Combination With Standard Therapy in Patients With Gastrointestinal Tumors
Brief Title: Evaluation of the Preliminary Efficacy and Safety of DR30206 in Combination With Standard Therapy in Patients With Gastrointestinal Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Zhejiang Doer Biologics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DR30206102
Record Dates: First submitted 2025-06-29; First posted 2025-07-09 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Gastrointestinal Cancer
Keywords: Gastrointestinal Cancer
MeSH Terms: conditions — Gastrointestinal Neoplasms | interventions — Oxaliplatin; Capecitabine; Leucovorin; Fluorouracil; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- DR30206+Oxaliplatin+Capecitabine (Experimental): DR30206 20mpk Q3W or DR30206 30mpk Q3W; Oxaliplatin 130 mg/m2, d1, Q3W; Capecitabine 1000 mg/m2, bid, d1-14, Q3W;
  Interventions: Drug: DR30206; Drug: Oxaliplatin; Drug: Capecitabine
- DR30206+Oxaliplatin+Calcium Folinate+5-FU (Experimental): DR30206 15mpk Q2W or DR30206 20mpk Q2W; Oxaliplatin 85 mg/m2, d1, Q2W; Calcium Folinate 400mg/m2, d1, Q2W; 5-FU 400mg/m2, d1 and 5-FU 1200mg/m2, d2-3, Q2W.
  Interventions: Drug: DR30206; Drug: Oxaliplatin; Drug: Calcium Folinate; Drug: 5-FU
- DR30206+Irinotecan+Calcium Folinate+5-FU (Experimental): DR30206 15mpk Q2W or DR30206 20mpk Q2W; Irinotecan 180 mg/m2, d1, Q2W; Calcium Folinate 400mg/m2, d1, Q2W; 5-FU 400mg/m2, d1 and 5-FU 1200mg/m2, d2-3, Q2W.
  Interventions: Drug: DR30206; Drug: Calcium Folinate; Drug: 5-FU; Drug: Irinotecan (CPT-11)

INTERVENTIONS:
Drug: DR30206 — Subjects receive DR30206 intravenously
Drug: Oxaliplatin — Subjects receive Oxaliplatin intravenously
  Arms: DR30206+Oxaliplatin+Calcium Folinate+5-FU; DR30206+Oxaliplatin+Capecitabine
Drug: Capecitabine — Subjects take Capecitabine orally
  Arms: DR30206+Oxaliplatin+Capecitabine
Drug: Calcium Folinate — Subjects receive Calcium Folinate intravenously
  Arms: DR30206+Irinotecan+Calcium Folinate+5-FU; DR30206+Oxaliplatin+Calcium Folinate+5-FU
Drug: 5-FU — Subjects receive 5-FU by Intravenous Bolus
  Arms: DR30206+Irinotecan+Calcium Folinate+5-FU; DR30206+Oxaliplatin+Calcium Folinate+5-FU
Drug: Irinotecan (CPT-11) — Subjects receive Irinotecan intravenously
  Arms: DR30206+Irinotecan+Calcium Folinate+5-FU

SUMMARY:
This is a multicenter, open-label phase Ib/IIa clinical study conducted in China, aimed at evaluating the safety tolerance, efficacy, pharmacokinetic (PK) characteristics, and immunogenicity of DR30206 in combination with standard treatment regimens for advanced or metastatic gastrointestinal tumors.

DETAILED DESCRIPTION:
This is a multicenter, open-label phase Ib/IIa clinical study conducted in China, aimed at evaluating the safety tolerance, efficacy, pharmacokinetic (PK) characteristics, and immunogenicity of DR30206 in combination with standard treatment regimens for advanced or metastatic gastrointestinal tumors.

The study consists of two phases: the dose escalation phase (phase Ib) and the dose expansion phase (phase IIa). Based on the tumor type and treatment approach of the participants, different cohorts are established within both the phases Ib and IIa.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign a written informed consent form.
2. Patients must be ≥ 18 and ≤75 years of age.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
4. Expected survival period of at least 3 months.
5. Depending on the tumor type, subjects must meet the following respective requirements:

   1. Colorectal cancer: i. Histologically or cytologically confirmed unresectable locally advanced or metastatic colorectal cancer; ii. Subjects who have not previously received systemic chemotherapy(except for left-sided colorectal cancer with wild-type RAS/BRAF); or subjects who have progressed after first-line chemotherapy with or without targeted or immunotherapy.
   2. Other gastrointestinal tumors: i. Histologically or cytologically confirmed unresectable locally advanced or metastatic esophageal adenocarcinoma, gastric adenocarcinoma, or gastroesophageal junction adenocarcinoma, with HER2-negative or low expression; ii. Subjects who have not previously received systemic chemotherapy; for patients who previously received adjuvant chemotherapy, neoadjuvant chemotherapy, or radical chemoradiotherapy for advanced disease with curative intent, if disease progression occurs more than 6 months after the completion of the last treatment, they are eligible for this study.
6. According to RECIST v1.1, subjects must have at least one measurable lesion.
7. Adequate bone marrow, liver, and renal function.
8. Male or female subjects with fertility must agree to take effective contraceptive measures during the study period and within 180 days after the end of the last medication.
9. Able to understand and follow the scheduled visits, treatments, laboratory tests, and other study procedures.

Exclusion Criteria:

1. Subjects with MSI-H or dMMR.
2. A history of severe allergic reactions to other monoclonal antibodies (mAb) or bispecific antibodies, or known allergies to any investigational drug or its components in this study.
3. Use of high-dose corticosteroids (>10 mg/day prednisone or equivalent doses of other corticosteroids) or other immunosuppressive drugs within 14 days prior to the first administration of the investigational drug.
4. Received the following treatments or medications within 28 days before starting the study treatment: a. Inoculate live attenuated vaccines, or expect to receive such vaccines during the study treatment period or within 5 months after the last administration of the study treatment; b.Systemic treatment with anti-tumor drugs, or local anti-tumor therapy.
5. Received local radiotherapy within 2 months prior to the first administration of investigational drug (palliative radiotherapy for bone metastasis completed more than 2 weeks before baseline tumor assessment is acceptable);
6. Received non-specific immunomodulatory therapy (e.g., interleukins, interferons, thymosin, tumor necrosis factor, etc.) within 2 weeks prior to the first administration of investigational drug;
7. Receipt of other investigational drugs or investigational medical devices within 28 days prior to the first administration of the investigational drug.
8. Major surgery (defined as requiring general anesthesia and hospitalization for more than 24 hours) or severe traumatic injury within 28 days prior to the first administration of the investigational drug, or expected to require major surgery during the study period, except for minor procedures (e.g., tooth extraction, biopsy) deemed not to affect participation in the study by the investigator.
9. Presence of severe chronic or active infections within 28 days prior to the first administration of the investigational drug, including but not limited to hospitalization for infection, sepsis, or severe pneumonia complications, or any active infection that the investigator considers may affect the participant's safety; or systemic antibiotic therapy within 2 weeks prior to the start of treatment (routine prophylactic anti-infective therapy is exempt).
10. Persistent clinically significant toxicities (CTCAE 5.0 Grade 2 or higher, e.g., hyperpigmentation, alopecia, etc.), except for adverse reactions deemed to have no safety risk by the investigator, related to prior treatments (including systemic therapy, radiotherapy, or surgery).
11. Presence of central nervous system (CNS) metastases and/or cancerous meningitis. Subjects who have received local treatment for brain metastases may be considered for participation in this study provided that imaging confirms no disease progression within 4 weeks prior to the first administration of the investigational drug, all neurological symptoms are stable, there is no evidence of new or enlarging CNS metastases, and radiotherapy, surgery, or corticosteroid therapy for CNS metastases has been discontinued for at least 28 days prior to the first administration of the investigational drug. However, cancerous meningitis, regardless of clinical stability, should be excluded.
12. Hepatitis B virus infection (must meet both HBsAg positive and HBV-DNA > 500 IU/mL), Hepatitis C virus infection (must meet both HCV-Ab positive and HCV-RNA positive), Human Immunodeficiency virus infection (HIV-Ab positive), active syphilis infection, active tuberculosis infection.
13. There have been clinically significant cardiovascular and cerebrovascular diseases within 6 months prior to the first study drug dosing.
14. Within 2 years prior to the first administration of the investigational drug, the subject has active autoimmune diseases requiring systemic treatment (e.g., use of glucocorticoids or immunosuppressive drugs). Replacement therapies (e.g., levothyroxine, insulin, or physiological corticosteroid replacement for adrenal or pituitary insufficiency) are permitted.
15. Within 3 years prior to the first administration of the investigational drug, the subject has a history of other malignancies, except those cured by definitive treatment with expectation of cure, such as basal or squamous cell skin cancer, localized low-risk prostate cancer, papillary thyroid cancer, or any in situ cancer treated by definitive resection (e.g., cervical intraepithelial neoplasia, ductal carcinoma in situ).
16. The subjects have other severe or uncontrolled medical conditions, or the investigator deems the subject unsuitable for participation in this clinical trial or believes it would affect the subject's adherence to the study protocol, including but not limited to: a) History of or current concomitant severe respiratory diseases; b) Severe arterial or venous thromboembolic events within 6 months prior to the first investigational drug administration; c) Massive pleural effusion, ascites, or pericardial effusion with clinical symptoms or requiring symptomatic treatment within 28 days prior to the first investigational drug administration; d) Active or history of inflammatory bowel disease; e) History of severe peptic ulcer, gastrointestinal perforation, fistula, gastrointestinal obstruction, intra-abdominal abscess, or acute gastrointestinal bleeding, or esophageal or gastric variceal bleeding due to portal hypertension within 6 months prior to the first investigational drug administration; f) History of clinically significant bleeding symptoms within 1 month prior to the first study drug administration; g) Imaging at screening shows tumor encasement of major vessels or presence of significant necrosis or cavitation, and the investigator judges that enrollment would increase the risk of bleeding.
17. The subject has a history of allogeneic hematopoietic stem cell transplantation or solid organ transplantation.
18. The subject has a history of substance abuse or a mental disorder that may affect compliance with the study.
19. Pregnant or breastfeeding women, where pregnancy is defined as the period from conception until the termination of pregnancy, and confirmed by a laboratory human chorionic gonadotropin (hCG) test within 7 days prior to the start of the study.
20. Other conditions deemed unsuitable for participation in this study by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2025-03-25 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Phase Ib: Incidence of dose limiting toxicities (DLTs) | 21 days or 28 days following first dose according to the arms.
  Dose-limiting describes side effects of a drug or other treatment that are serious enough to prevent an increase in dose or level of that treatment.
Phase Ib: Incidence and severity of treatment-emergent adverse events (TEAEs) | From the first dose up to 90 days after the last dose or initiation of new anti-tumor treatment
  The incidence and severity of AEs graded according to NCI-CTCAE v5.0.
Phase Ib: Maximum tolerated dose(MTD) | 21 days or 28 days following first dose according to the arms.
  As measured by number of participants experiencing dose related toxicity (DLT) in each escalating cohort.
Phase Ib: Recommended phase 2 dose (RP2D) | 21 days or 28 days following first dose according to the arms.
  A recommended phase 2 dose will be determined based on safety data.
Phase IIa: Objective response rate (ORR) (RECIST v1.1) of DR30206 in combination with standard therapy for the treatment of other gastrointestinal tumors | the period from the date of initial medication to the objective recording of disease progression according to RECIST 1.1 standards or to the start of new anti-tumor treatment (whichever occurs first)
  Objective response rate (ORR) is the proportion of subjects with complete response (CR) or partial response (PR), based on RECIST v1.1
Phase IIa: Objective response rate (ORR) (RECIST v1.1) of DR30206 in combination with standard therapy for the treatment of advanced or metastatic colorectal cancer. | the period from the date of initial medication to the objective recording of disease progression according to RECIST 1.1 standards or to the start of new anti-tumor treatment (whichever occurs first), assessed up to 24 months
  Objective response rate (ORR) is the proportion of subjects with complete response (CR) or partial response (PR), based on RECIST v1.1

CONTACTS AND LOCATIONS:
Overall Officials: Yanshan Huang CEO, Study Chair — Zhejiang Doer Biologics Co., Ltd.; Ruihua Xu, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China